CLINICAL TRIAL: NCT03862092
Title: Frequency of Putative Enteric Zoster Diagnosed Using Saliva Samples in Patients With Abdominal Pain: a Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Han Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-1186
Record Dates: First submitted 2019-03-02; First posted 2019-03-05 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Abdominal Pain; Zoster With Other Complications
Keywords: varicella zoster virus; enteric zoster; saliva
MeSH Terms: conditions — Abdominal Pain; Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with acute abdominal pain (Experimental): Salivary VZV-DNA PCR was performed in patients who visited the emergency room due to acute abdominal pain.
  Interventions: Diagnostic Test: Salivary VZV-DNA PCR

INTERVENTIONS:
Diagnostic Test: Salivary VZV-DNA PCR — VZV-DNA PCR of saliva samples

SUMMARY:
The aim of this study is to identify the frequency of enteric zoster using salivary varicella zoster virus (VZV) DNA PCR in patients who visit the emergency room due to acute abdominal pain.

DETAILED DESCRIPTION:
Varicella zoster virus (VZV) infects and establishes latency in neurons in the ganglia of the cranial nerve, dorsal root, and enteric ganglia. VZV reactivation in enteric neurons (enteric zoster) can cause nonspecific abdominal pain and/or serious gastrointestinal dysfunction without cutaneous manifestations. Detection of VZV DNA in saliva may be useful for identifying enteric zoster. We evaluated the frequency of putative enteric zoster based on the presence of salivary VZV DNA in patients with acute abdominal pain.

Adult patients who visited the emergency room due to moderate to severe acute abdominal pain were prospectively enrolled at a tertiary hospital between May 2019 and November 2019. Abdominopelvic computed tomography (APCT) was performed in all patients. Saliva samples were collected from all studied patients. Enteric zoster was suspected based on the presence of salivary VZV DNA, detected using real-time polymerase chain reaction (PCR).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18, and < 80 years
* ER-visited patients with acute abdominal pain

  * Numerical rating scale (NRS) score ≥ 4
  * Unresponsive to gastrointestinal motility drug, antacid

Exclusion Criteria:

* Unwilling or unable to give informed consent forms
* Patients taking antiviral agents
* Patients complaining mild abdominal pain (NRS score ≤ 3)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of enteric zoster in patients with acute abdominal pain | At the time of enrolled.
  The frequency of putative enteric zoster in patients with acute abdominal pain regardless of their underlying diseases

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Han Kim, MD.PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zerboni L, Sen N, Oliver SL, Arvin AM. Molecular mechanisms of varicella zoster virus pathogenesis. Nat Rev Microbiol. 2014 Mar;12(3):197-210. doi: 10.1038/nrmicro3215. Epub 2014 Feb 10. PMID 24509782
- [Background] Dworkin RH, Johnson RW, Breuer J, Gnann JW, Levin MJ, Backonja M, Betts RF, Gershon AA, Haanpaa ML, McKendrick MW, Nurmikko TJ, Oaklander AL, Oxman MN, Pavan-Langston D, Petersen KL, Rowbotham MC, Schmader KE, Stacey BR, Tyring SK, van Wijck AJ, Wallace MS, Wassilew SW, Whitley RJ. Recommendations for the management of herpes zoster. Clin Infect Dis. 2007 Jan 1;44 Suppl 1:S1-26. doi: 10.1086/510206. PMID 17143845
- [Background] Gilden DH, Kleinschmidt-DeMasters BK, LaGuardia JJ, Mahalingam R, Cohrs RJ. Neurologic complications of the reactivation of varicella-zoster virus. N Engl J Med. 2000 Mar 2;342(9):635-45. doi: 10.1056/NEJM200003023420906. No abstract available. PMID 10699164
- [Background] Gilden DH, Wright RR, Schneck SA, Gwaltney JM Jr, Mahalingam R. Zoster sine herpete, a clinical variant. Ann Neurol. 1994 May;35(5):530-3. doi: 10.1002/ana.410350505. PMID 8179298
- [Background] Edelman DA, Antaki F, Basson MD, Salwen WA, Gruber SA, Losanoff JE. Ogilvie syndrome and herpes zoster: case report and review of the literature. J Emerg Med. 2010 Nov;39(5):696-700. doi: 10.1016/j.jemermed.2009.02.010. Epub 2009 Mar 27. PMID 19327938
- [Background] Gershon AA, Gershon MD. Pathogenesis and current approaches to control of varicella-zoster virus infections. Clin Microbiol Rev. 2013 Oct;26(4):728-43. doi: 10.1128/CMR.00052-13. PMID 24092852
- [Background] Mehta SK, Tyring SK, Gilden DH, Cohrs RJ, Leal MJ, Castro VA, Feiveson AH, Ott CM, Pierson DL. Varicella-zoster virus in the saliva of patients with herpes zoster. J Infect Dis. 2008 Mar 1;197(5):654-7. doi: 10.1086/527420. PMID 18260763
- [Background] Park SY, Kim JY, Kim JA, Kwon JS, Kim SM, Jeon NY, Kim MC, Chong YP, Lee SO, Choi SH, Kim YS, Woo JH, Kim SH. Diagnostic Usefulness of Varicella-Zoster Virus Real-Time Polymerase Chain Reaction Analysis of DNA in Saliva and Plasma Specimens From Patients With Herpes Zoster. J Infect Dis. 2017 Dec 27;217(1):51-57. doi: 10.1093/infdis/jix508. PMID 29029120
- [Derived] Ra SH, Kwon JS, Kim JY, Cha HH, Lee HJ, Jung J, Kim MJ, Chong YP, Lee SO, Choi SH, Kim YS, Kim WY, Kim SH. Frequency of putative enteric zoster diagnosed using saliva samples in patients with abdominal pain: a prospective study. Infect Dis (Lond). 2021 Sep;53(9):713-718. doi: 10.1080/23744235.2021.1908593. Epub 2021 Apr 8. PMID 33830871